CLINICAL TRIAL: NCT07199894
Title: A Randomized Controlled Trial Comparing Mirabegron and Solifenacin Combination Therapy Versus Desmopressin Monotherapy in Treatment of Children With Primary Mono-Symptomatic Nocturnal Enuresis
Brief Title: Omegapres Versus Solifenacin and Mirabegron Combination Therapy in Treatment of Primary MNE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.24.07.2820
Record Dates: First submitted 2025-08-18; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Nocturnal Enuresis in Children
Keywords: nocturnal enuresis; Desmopressin; Mirabegron; Solifenacin; B3 agonist; Anti-cholinergic; Randomised controlled trial
MeSH Terms: conditions — Nocturnal Enuresis | interventions — mirabegron; Cholinergic Antagonists; Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADH analougue monotherapy (Sham Comparator): Desmopressin
  Interventions: Drug: Desmopressin (DDAVP)
- Anticholinergic and b3 agonist combination (Experimental): Solifenacin and Mirabegron
  Interventions: Drug: Mirabegron (beta3-adrenoceptor agonist), Anticholinergics

INTERVENTIONS:
Drug: Mirabegron (beta3-adrenoceptor agonist), Anticholinergics — Anticholinergic and B3 agonist drugs used for treatment of mono-symptomatic nocturnal enuresis
  Arms: Anticholinergic and b3 agonist combination
Drug: Desmopressin (DDAVP) — ADH analogue in treatment of mono-symptomatic nocturnal enuresis
  Arms: ADH analougue monotherapy

SUMMARY:
The goal of this clinical trial is to compare combination of Solifenacin and MIrabegron in treatment of primary mono-symptomatic nocturnal enuresis in children. It will also learn about the safety of that combination. The main questions it aims to answer are:

Does combination of Solifenacin and MIrabegron lower the number of wet nights? What medical problems do participants have when taking combination of Solifenacin and MIrabegron? Researchers will compare the combination to omegapress to see if the combination works better to treat primary mono-symptomatic nocturnal enuresis.

Participants will:

Take the combination or Omegapress every day for 3 months Visit the clinic once monthly for checkups and tests Keep a diary of their symptoms and the number of wet nights

DETAILED DESCRIPTION:
Nocturnal enuresis (NE) is defined as intermittent incontinence during sleep in a child aged 5 years or more in the absence of congenital anomalies of the urinary tract or congenital or acquired defects of the central nervous system. It affects 15-20% of children aged 5 years and 1-2% of adolescents with spontaneous recovery occurs at a rate of 10-15% per year. About 75% of affected children have primary nocturnal enuresis, who never attained continence for longer than 6 months during sleep. Patients with mono-symptomatic nocturnal enuresis (MNE) do not have any other symptoms of lower urinary tract dysfunction.

The standard view of NE pathogenesis as being the result of either nocturnal polyuria or nocturnal detrusal overactivity with high arousal thresholds has become well-established, but further research now complicates the picture. First, Psychological/psychiatric problems are overrepresented in enuresis and might in a minority of cases have a causal or aggravating role. Second, Nocturnal polyuria is not always linked to vasopressin deficiency. Third, nocturnal detrusal overactivity is in itself pathogenetically heterogeneous, and could be linked to constipation. Fourth, Sleep of enuretic children might be "deep," but possibly also disturbed (by obstructed airways or a distended or contracting bladder).

Standard first line treatments for MNE are alarm therapy or desmopressin. Alarm therapy conditions the child to inhibit urination during sleep or to wake to void when the bladder is full. Desmopressin decreases the amount of overnight urine produced, thereby reducing the need to wake to void. Tricyclic antidepressants are also sometimes used for treating enuresis.

Combination therapy of desmopressin plus alarm is often taken into consideration when the patients are refractory to single treatment, have behavioral problems or frequent night-time enuresis. Anticholinergic agents (AA), such as tolterodine, oxybutynin and propiverine, can prevent involuntary detrusal contractions. They can significantly decrease urge incontinence in children. Desmopressin plus AA therapy is often used in non-responders to desmopressin monotherapy or in those with a restricted bladder capacity and thickened bladder wall.

Desmopressin is more effective and has lower rate of side effects in comparison to Oxybutynin for treatment of NE. However, it has been proved that desmopressin plus AA combination (Oxybutynin or Solifenacin) therapy has higher response rates and lower relapse rates compared with desmopressin monotherapy as first-line treatment for children with primary mono-symptomatic nocturnal enuresis (PMNE) with an acceptable tolerability profile. This can be explained by bladder reservoir dysfunction during sleep which is relatively common in MNE. This phenomenon may explain treatment failure with desmopressin, despite adequate antidiuretic response. In combination therapy, desmopressin reduces urine production and the AA allows the bladder to store more urine due to increased functional bladder capacity.

Adrenoceptors have two main groups, α and β, and several subtypes. β1-, 2- and 3-adrenoceptors have been identified in human urothelium and detrusor muscle, with β3 being highly expressed in the urinary bladder. β3-adrenoceptors have been demonstrated as the predominant subtype, with 95% of all β-adrenoceptor mRNA in the human bladder relating to this subtype; this receptor is thought to be important for mediating human detrusal relaxation. This is supported by animal studies in which β3-adrenoceptor agonists have been demonstrated to cause dose-dependent detrusal relaxation during the storage phase of the micturition cycle and to inhibit neurogenic detrusal overactivity during in vitro studies. Mirabegron, a β3-adrenoceptor agonist, improves storage function and subjective symptoms without affecting voiding function in women with OAB.

To the best of our knowledge, no study used AA plus Mirabegron for treatment of PMNE In this study, we hypothesize that the combined detrusal relaxing effect of AA and β3- adrenoceptor agonist will produce better outcome regarding number of wet nights than desmopressin monotherapy in children with PMNE.

ELIGIBILITY:
Inclusion Criteria:

Primary mono-symptomatic nocturnal enuresis -

Exclusion Criteria:

Bowel dysfunction Psychatric illness Respiratory sleep disorders

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of improvement in number of wet nights per week | 90 days
  Counting number of wet nights per week before and after receiving treatment and the resulting percentage will be the primary end point.

SECONDARY OUTCOMES:
Number of patients who experienced side effects in response to each treatment. | 90 days
  Each patient will be followed up monthly during the 3 months period and surveyed for side effects. The number of patients who experienced side effects will be compared between the two groups and compare the number of patients who subsequently discontinued the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology center - Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol